CLINICAL TRIAL: NCT00212589
Title: A Randomized Crossover Trial Comparing Oral Capecitabine and Intravenous Fluorouracil + Folinic Acid (Nordic FU/FA Regimen) for Patient Preference in Colorectal Cancer
Brief Title: Patients Preference for Oral or i.v. Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 11.02
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2005-09-21 (Estimated); Status verified 2004-05

CONDITIONS: Colorectal Cancer
Keywords: Patients preference; Colorectal cancer; Capecitabine; Fluorouracil + folinic acid; Cross-over study
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Capecitabine; Fluorouracil; Leucovorin

INTERVENTIONS:
Drug: Capecitabine
Drug: Fluorouracil + folinic acid

SUMMARY:
Until recently, bolus 5-flourouracil (FU) + folinic acid (FA) has been considered the standard chemotherapy for patients with colorectal cancer. Several studies have shown that Capecitabine is as effective as Mayo regimen. The Nordic FU/FA schedule was developed to be an active and tolerable bolus regimen. The Nordic regimen consists of a short (3 minutes) bolus injection of FU and 30 minutes later FA for 2 consecutive days each 2 weeks. In randomized studies efficacy is comparable to other FU/FA regimens.

It is claimed that patients prefer oral therapy and in a randomized study comparing oral therapy (UFT/FA) and bolus FU/FA (Mayo) 84% preferred oral therapy.

In the present randomized cross-over study patients were randomized for 3 courses of Nordic FU/FA followed by 2 courses of Capecitabine (or vice versa), and patients were asked for their preference.

ELIGIBILITY:
Inclusion Criteria:

* Indication for treatment with a FU-regime
* WHO Performance Status 0-1
* Life expectancy > 3 months
* Adequate haematological, renal and hepatic functions
* Adequate contraceptives
* Written informed consent

Exclusion Criteria:

* Known CNS-metastases
* Prior treatment with chemotherapy
* Pregnant or breast feeding women
* Current infection, unresolved bowel obstruction or subobstruction, uncontrolled Crohn's disease or ulcerative colitis
* other serious illness or medical conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2002-12; Study Completion 2004-04

CONTACTS AND LOCATIONS:
Overall Officials: Per Pfeiffer, MD, Principal Investigator — Department of Oncology, Odense University Hospital, DK-5000 Odense C, Denmark
Locations (4):
- Denmark (4):
  - Department of Oncology, Esbjerg Hospital, Esbjerg
  - Department of Oncology, Odense University Hospital, Odense
  - Department of Oncology, Sonderborg Hospital, Sønderborg
  - Department of Oncology, Vejle Hospital, Vejle

REFERENCES:
- [Background] Lima AP, del Giglio A. Randomized crossover trial of intravenous 5-FU versus oral UFT both modulated by leucovorin: a one-centre experience. Eur J Cancer Care (Engl). 2005 May;14(2):151-4. doi: 10.1111/j.1365-2354.2005.00531.x. PMID 15842464
- [Background] Borner MM, Schoffski P, de Wit R, Caponigro F, Comella G, Sulkes A, Greim G, Peters GJ, van der Born K, Wanders J, de Boer RF, Martin C, Fumoleau P. Patient preference and pharmacokinetics of oral modulated UFT versus intravenous fluorouracil and leucovorin: a randomised crossover trial in advanced colorectal cancer. Eur J Cancer. 2002 Feb;38(3):349-58. doi: 10.1016/s0959-8049(01)00371-9. PMID 11818199